CLINICAL TRIAL: NCT05676658
Title: Effects of Coherent Breathing Breathwork on Mental Health and Wellbeing: A Randomised Placebo-controlled Study
Brief Title: Effects of Coherent Breathing Breathwork on Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Collaborators: Sylff Association (Unknown)
Responsible Party: Principal Investigator, Guy Fincham, Guy William Fincham, University of Sussex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sussex coherent breath study
Record Dates: First submitted 2022-12-14; First posted 2023-01-09 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Stress; Anxiety; Depressive Symptoms; Wellbeing; Sleep Disturbance
MeSH Terms: conditions — Anxiety Disorders; Depression; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coherent breathing (Experimental)
  Interventions: Behavioral: Coherent breathing
- Placebo coherent breathing (Placebo Comparator)
  Interventions: Behavioral: Placebo coherent breathing

INTERVENTIONS:
Behavioral: Coherent breathing — Guided audio of coherent breathing pre-recorded by trained breathwork facilitator: ~5.5bcpm (with equal inhalation/exhalation durations of ~5.5secs each) for ~10mins/day over four weeks / 28 days. Delivered remotely through audio link.
  Arms: Coherent breathing
Behavioral: Placebo coherent breathing — Same audio of coherent breathing but paced at: ~12bcpm (with equal inhalation/exhalation durations of 2.5secs each) for ~10mins/day over four weeks / 28 days.
  Arms: Placebo coherent breathing

SUMMARY:
The investigators are conducting a randomised-controlled trial comparing coherent breathing at ~5.5 breath cycles per minute-bcpm (with equal inhalation/exhalation durations of ~5.5secs each) to a well-designed placebo (paced breathing at 12bcpm with equal inhalation/exhalation durations of 2.5secs each). The metric of 12bcpm is in line with guidance from the British Journal of Nursing, Royal College of Physicians, and Johns Hopkins University which state that the average, healthy bcpm should range from: 12-20bcpm, 12-18bcpm, and 12-16bcpm, respectively, hence the investigators chose the minimum/lower bound for the active placebo control group. The main questions that our study attempts to address are: Does coherent breathing (and placebo coherent breathing) lead to improved mental health and wellbeing in a general population adult sample?

The study will be conducted entirely online through the research platform Prolific, so participant data will be anonymous. The investigators will collect self-reports of mental health and wellbeing before and after the four-week breathwork period, along with a follow-up one-month later. Pre-post intervention and follow-up questionnaires will be completed online via the survey platform Qualtrics which will be linked to Prolific. Participants will also be asked how many times they practiced out of the assigned 28 days, to gauge self-reported adherence to the protocol. The investigators can then observe whether self-reported adherence correlates with changes in mental health and wellbeing, if any. Data on the self-reported credibility/expectancy of the breathwork randomly allocated to participants will also be collected, along with open-ended responses on participants' overall experience of the protocol/study.

ELIGIBILITY:
Inclusion Criteria (self-assessed):

* 18+ years of age (18 is the automatic minimum age on Prolific)
* Able to breathe through nose
* Have access to headphones
* The following pre-screeners on Prolific will also be set so only those eligible on Prolific will see the study: Located/living in UK, Fluent in English, approval rate of 98% and at least 20 previous submissions (as recommended by Prolific to increase retention and reduce dropout rates in longitudinal and multi-part studies)

Exclusion Criteria (self-assessed):

* Any problems which affect ones ability to pace their breathing (i.e., active/chronic respiratory infection including blocked nose/cough/cold/fever, etc.), breathlessness, cardiovascular problems, respiratory conditions or diseases (i.e., uncontrolled symptomatic asthma, COPD, lung cancer, etc.), abnormally slow breathing (bradypnea), or abnormally fast breathing (tachypnoea)
* Any other physical/mental health conditions or current life events which impair or affect ones ability to engage in activities involving breath control

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Subjective stress | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and four weeks after the intervention). Primary timepoint is post-intervention
  Depression Anxiety Stress Scale-21 (DASS-21) - stress subscale (score range: 0-21; higher scores denote worse outcome). Score on DASS-21 is then multiplied by two to convert it to the longer form DASS-42 final score

SECONDARY OUTCOMES:
Subjective anxiety | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and four weeks after the intervention)
  DASS-21 - anxiety subscale (score range: 0-21; higher scores denote worse outcome)
Subjective depressive symptoms | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and four weeks after the intervention)
  DASS-21 - depression subscale (score range: 0-21; higher scores denote worse outcome)
Subjective wellbeing | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and four weeks after the intervention)
  The World Health Organisation-5 Well-Being Index (WHO-5) (score range: 0-25; higher scores denote better outcome)
Subjective sleep disturbance | Pre-post intervention and follow-up (immediately before the intervention, immediately after the intervention, and four weeks after the intervention)
  PROMIS Item Bank v1.0 - Sleep Disturbance - Short Form 8a (score range: 5-40; higher scores denote worse outcome). Data scored using a T-score transformation according to PROMIS Sleep scoring manual on: www.healthmeasures.net
Self-reported adherence to protocol | Post-intervention (immediately after the intervention)
  Number of sessions participants self-report practicing out of 28 days assigned
Self-reported credibility and expectancy of protocol | Immediately after starting breathwork intervention
  Credibility/Expectancy Questionnaire (CEQ-6). Two Sets (Credibility of course/therapy [breathwork] and expectancy of course/therapy [breathwork]). Four items scored 1-9 and two items scored 0-100%. Higher scores denote greater credibility and/or expectancy of specific breathwork technique

OTHER OUTCOMES:
Overall experience | Post-intervention and follow-up (immediately after the intervention, and four weeks after the intervention)
  Optional open-ended questions on participants' perspectives and overall experience of the protocol/study-period
Impairment of practice | Post-intervention (immediately after the intervention)
  Optional open-ended question on whether anything impaired participants' ability to perform their randomly allocated breathwork
Hypothesis guessing | Follow-up (four weeks after the intervention)
  Optional open-ended question on whether participants can guess the hypothesis of the study

CONTACTS AND LOCATIONS:
Overall Officials: Guy W Fincham, MSc, Principal Investigator — University of Sussex
Locations (1):
- Prolific, Remote/Online, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All participant data will be anonymous (only Prolific user IDs will be seen). No identifiable personal information will be collected. Participants will be able to check a box if they are happy for our research team at the University of Sussex to include the data again in future studies related to breathwork and meditation if these have gained independent ethically approval, based on the strict confidentiality terms described in the participant info/consent form.
Time Frame: Indefinitely after the study has been completed.
Access Criteria: Our research team at the University of Sussex will have access. The datasets used and/or analysed during the current study will be available from the principal investigator on reasonable request to other researchers working on meditation and breathwork.

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05676658/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05676658/SAP_001.pdf